CLINICAL TRIAL: NCT05173701
Title: Effects of Probiotics on Peripheral Immunity in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Franca Marino (Other)
Collaborators: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other); Università degli Studi dell'Insubria (Other)
Responsible Party: Sponsor-Investigator, Franca Marino, Professor, Università degli Studi dell'Insubria
Organization: Università degli Studi dell'Insubria (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PROB-PD
Record Dates: First submitted 2021-11-08; First posted 2021-12-30 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Probiotics; Immunomodulation; Microbiota
MeSH Terms: conditions — Parkinson Disease | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Administration of a mixture of probiotics once daily for three months
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Administration of a placebo (maltodextrin) once daily for three months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Selected probiotics mixture, in powder form, will be administered once daily for three months in the morning.
  Arms: Probiotics
Dietary Supplement: Placebo — A placebo (2,7g maltodextrin) will be administered once daily for three months in the morning.
  Arms: Placebo

SUMMARY:
Parkinson's Disease (PD) is a common neurodegenerative disease, with no disease-modifying treatment available, therapy is therefore only symptomatic. The pathophysiology of the disease is still unclear, but inflammatory mechanisms are reported to play a prominent role. An involvement of peripheral adaptive immunity, with an imbalance in T cell subpopulations and in the expression of transcriptional factors (TF) in Cluster of Differentiation (CD) 4 positive T cells has been reported. An initial aggregation of α-synuclein (α-syn) in the gut with subsequent propagation along the vagus nerve to the brain has also been hypothesised. Interestingly, in an α-syn overexpressing murine model, the absence of gut microbiota prevented both microglia activation and motor impairment, pointing to a fundamental role of the microbiota in the development of PD. It has been shown that in Peripheral Blood Mononuclear Cells (PBMC) of PD patients, probiotics modulate the in vitro production of cytokines toward an anti-inflammatory profile. The investigators developed a clinical trial protocol for the evaluation of probiotics' effects on the peripheral immune system profile in Parkinson's Disease patients. ROS, Lymphocyte subpopulations, TF levels in PBMC will be assessed at baseline and after treatment with a mixture of probiotics in PD patients to assess immunomodulatory effects of said treatment. Motor and non-motor symptoms of PD will also be monitored through the trial period.

DETAILED DESCRIPTION:
Introduction Parkinson's Disease (PD) is a common neurodegenerative disease, affecting up to 1-2 people in 1000 at any given time. Prevalence increases with age and is estimated at 1% in people over 65.

There is no available treatment to prevent PD onset or to delay its progression and therapy is focused on symptoms management. The administration of carbidopa/levodopa allows for control of motor symptoms, but it becomes less effective as the disease progresses and increasing daily doses causes more frequent and severe side effects.

The histopathologic hallmark of PD is the loss of dopaminergic neurons and accumulation of α-synuclein (α-syn) in surviving neurons, but the underlying pathophysiology is still unclear. Inflammatory mechanisms have been suggested to play a prominent role in the disease, with an imbalance between detrimental and protective immune functions, as well as neurotoxicity caused by reactive oxygen species (ROS).

Further evidence highlights the involvement of peripheral adaptive immunity in PD, reporting an imbalance in T cell subpopulations and in the expression of transcriptional factors in CD4+ T cells in PD patients.

In these patients, non-motor symptoms may precede the onset of a clinically established disease.

Etiopathogenesis of PD is still unknown, but seminal work by Braak et al. hypothesised an initial aggregation of α-syn in the gut with subsequent propagation along the vagus nerve to the brain, finally reaching the substantia nigra in the mesencephalon.

Interestingly, in an α-syn overexpressing murine model of PD, the absence of gut microbiota prevented both microglia activation and motor impairment, thus pointing to a fundamental role of the gut and microbiota in the pathogenesis and development of PD.

In a recent paper, Magistrelli et al. confirmed that probiotics may influence the peripheral immune system. Particularly, in peripheral blood mononuclear cells (PMBCs) of a cohort of PD patients, probiotics were able to modulate the production of cytokines toward an anti-inflammatory profile and to reduce the production of reactive oxygen species (ROS). The clinical effects of probiotics have been also explored in other pathological conditions. Tankou et al. administered VSL#3 in a cohort of 9 multiple sclerosis patients, whose peripheral immune system shifted toward an anti-inflammatory profile, with an inverse tendency after VSL#3 discontinuation. These results were also confirmed by the same group after administration of a mix of probiotics (four strains of Lactobacillus and three strains of Bifidobacterium).

In the light of this evidence, the investigators designed a randomised controlled clinical trial whose primary objective is to test whether probiotics can influence the peripheral immune system in a cohort of PD patients. The aim of the protocol is to highlight changes in transcriptional factors messenger Ribonucleic Acid (mRNA) levels, lymphocytes subpopulations (Th1, Th2, Th17 and Treg), cytokine levels and ROS production.

Methods and analyses This explorative study is a randomized placebo-controlled double-blind study to evaluate the efficacy of probiotics in modulating the peripheral immune system in Parkinson's Disease subjects. Participants will be randomised in two comparable groups and treated with a mixture of probiotics or matching placebo once daily for three months. The primary objective of this study is to verify the effects of probiotics on the peripheral immune system. As exploratory outcomes, motor and non-motor symptoms of PD will be monitored, as well as cognitive function and quality of life over the three months treatment period via a selection of clinical rating scales.

Participant identification Subjects will be recruited among patients with scheduled routine follow-up visits at Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara. Detailed information on comorbidities, current medical therapy and demographic data of these subjects will be readily available. The trial design will be briefly outlined and patients will be asked about their interest in participating. Willing subjects will attend a screening visit, written informed consent will be obtained before confirming eligibility.

Trial procedures

Clinical During enrolment visit, medical and neurological examination will assess the need for immediate variations in medical therapy for each participant. Within two weeks, any therapy modification will be completed and baseline visit will be scheduled.

During baseline visit (T0), physical and neurological examinations will be repeated to confirm the subject's conditions and persistence of inclusion criteria, a baseline blood withdrawal will be performed and all clinical evaluation scales will be completed to set baseline scores. Each participant, after the subscription of an appropriate informed consent, will be randomized and given a treatment box, containing single-dose sachets with 2,7g of powder of the allocated formulation. Patients will be instructed to take daily doses at home every morning before breakfast, mixing the content of one sachet in about 125 ml of fresh water or other cold, non-carbonated drink. Participants will be instructed to keep unused or empty packaging for recollection and compliance evaluation.

Follow-up visits will be scheduled at 4 weeks after T0 (T1) and at 12 weeks after T0 (T2). At T1, physical and neurological examination will be repeated and all clinical scales administered again. At T2, all assessments performed at T0 will be carried out again, including blood withdrawal.

At T0 and T2, withdrawal of 40 ml venous blood will be performed after a fasting night, between 8:00 and 10:00 am, in ethylenediaminetetraacetic acid-coated tubes (BD Vacutainer). Tubes will be coded and stored at room temperature until processing, within 24 hours. Complete blood count with differential analysis will be conducted on separate blood samples.

Laboratory methods

Cytokine measurement The possible influence of probiotic treatment on inflammatory profile will be evaluated by measuring at T0 and T2 the plasma levels of pro (e.g. Tumor Necrosis Factor (TNF)-α, Interferon (IFN)-γ) and anti-inflammatory cytokines (Interleukin (IL)-10, IL-4). Plasma aliquots from every sample will be separated and stored for cytokines assays. 2 mL of fresh blood will be centrifuged at 1400g for 10 minutes at room temperature and two plasma aliquots of 350 µL each will be stored in 1,5mL vials to assay cytokines levels.

Flow cytometric evaluation of immune phenotype In order to investigate possible changes in immune phenotype, the profile of both innate and adaptive immunity will be deepened by means of a cytofluorimetric evaluation according to the strategy described by Kustrimovic et al. in 2018 and with additional panels aimed specifically dedicated to innate immunity. The following cell subsets of the adaptive immune system will be assessed: CD4+ and CD8+ T naïve/memory cells, CD4+ T helper subsets and CD4+ regulatory T cells. Moreover, for innate immunity, monocytes and Natural Killer (NK) cells will be also assessed. Acquisition will be performed on a BD Fluorescence-activated cell sorting (FACS) Celesta flow cytometer (Becton Dickinson Italy, Milan, Italy) with BD FACS Diva software (version 8.0.1.1) and data will be analysed with FlowJo software (version 10.7.1)

Transcriptional factors mRNA evaluation According to previous studies by Kustrimovic and De Francesco, the ability of probiotic treatment to modify mRNA levels of the main transcriptional factors in CD4+ T lymphocytes will also be investigated. CD4+ positive cells will be obtained by PBMC, which will be isolated from whole blood using Ficoll-Paque Plus density gradient centrifugation. After resuspension, residual contaminating erythrocytes will be lysed by addition of 10 mL of lysis buffer ((g/L) NH4Cl 8.248, KHCO3 1.0, EDTA 0.0368). Cells will be washed twice in Purified Bovine Serum (PBS) by addition of 10 mL of PBS, then centrifuged at 300 g for 10 min at room temperature and resuspended in 10 mL of Roswell Park Memorial Institute medium (RPMI)/10% Fetal Bovine Serum (FBS). Manual cell count will then be performed to set CD4 separation reagents quantities.

Typical PBMC preparations will contain at least 80% lymphocytes. CD4+ T cells will then be isolated from PBMC by means of Dynabeads CD4 Positive Isolation kit. At least 50,000 separated CD4+ T cells will then be resuspended in PerfectPure RNA lysis buffer (5 Prime GmbH, Hamburg, Germany), and total RNA will be extracted by PerfectPure RNA Cell Kit™.

Reverse-transcription will be performed on resulting mRNA using a random primer and a high-capacity complementary DNA (cDNA) Real Time (RT) kit.

RT-Polymerase Chain Reactions (PCR) will be performed with 1 μM cDNA. Amplification of cDNA will allow for the analysis of mRNA levels of the transcription factor genes TBX21, STAT1, STAT3, STAT4, STAT6, RORC, GATA3, FOXP3 and NR4A2.

Treatment composition and rationale

Treatment:

Bifidobacterium animalis subsp. lactis BS01 ≥ 1 x 10^9 Colony Forming Units (CFU) Bifidobacterium longum 03 ≥ 1 x 10^9 CFU Bifidobacterium adolescentis BA02 ≥ 1 x 10^9 CFU Fructo-oligosaccharides FOS 2500 mg Maltodextrin q.s.

Placebo:

Maltodextrin q.s.

Each probiotics formulation contains Bifidobacterium animalis subsp. lactis (BS01), Bifidobacterium longum (BL03) and Bifidobacterium adolescentis (BA02). Fructo-oligosaccharides (FOS) is added as a prebiotical component and maltodextrin is used as a bulking agent.

The choice of probiotics for this study is based on solid literature data: in particular PBMC of PD patients treated with Bifidobacterium animalis subsp. Lactis (BS01) showed an increased production of anti-inflammatory cytokine IL-10. Said treatment also supported restoration of membrane integrity in a model of CacO2-cells.

All probiotics used are included in the "Qualified Presumption of Safety (QPS)-recommended biological agents intentionally added to food or feed as notified to European Food Safety Authority (EFSA) 12".

The placebo formulation is solely composed by maltodextrin.

Sample size calculation, data analysis The design of this study is explorative and equally randomised to treatment with probiotics or placebo. Due to the exploratory nature of the proposed study, a formal sample size calculation is not strictly required. Sample size for this study has thus been based mainly on previous results from another in vitro study, which yielded statistically significant results in a small cohort of 40 PD patients for all tested probiotic strains, with a global reduction in proinflammatory cytokines production and an increase in anti-inflammatory cytokines. In the present study, the expected sample will be doubled, with a total of 80 specimens to be collected both at T0 and T2.

Data from previous in vitro study has been used to estimate orientational sample sizes for the in vitro effect of all tested probiotic strains and a sample size of 80 subjects allows for the determination of most tested cytokines variations with an expected power greater than 80%, setting the threshold for statistical significance at 0.05.

Statistical analysis on collected data will be performed after assessing normality of data distribution and using two-tailed Student's t test or Mann-Whitney test as appropriate for independent variables comparisons. Data correlations will be analysed through Pearson's or Spearman's correlation tests. ANOVA or the Kruskal-Wallis tests will be used for comparisons between more than two groups and paired t-test or Wilcoxon signed ranks test will be used when comparing paired groups (e.g. baseline vs end of treatment, treatment vs placebo). Thresholds for statistical significance will be set according to the specific test characteristics.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of Parkinson's Disease;
* a disease duration between 2 and 5 years at baseline

Exclusion Criteria:

* past or concomitant autoimmune disease
* previous or ongoing immune-modulating or immunosuppressive therapy
* inflammatory bowel diseases, colorectal diseases or past major abdominal or pelvic surgery
* antibiotics therapy up to three months before enrolment
* usage of tube feeding
* known or suspected allergy to any component of the treatment or placebo mixtures
* known and established cognitive decline or any comorbidity preventing reliable completion of trial assessments
* motor fluctuations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma IFN-γ level | Baseline, 12 weeks
  IFN-γ level will be assessed in plasma samples via ELISA assay.
Changes in plasma TNF-α level | Baseline, 12 weeks
  TNF-α level will be assessed in plasma samples via ELISA assay.
Changes in plasma IL-4 level | Baseline, 12 weeks
  IL-4 level will be assessed in plasma samples via ELISA assay.
Changes in plasma IL-17A level | Baseline, 12 weeks
  IL-17A level will be assessed in plasma samples via ELISA assay.
Changes in plasma IL-10 level | Baseline, 12 weeks
  IL-10 level will be assessed in plasma samples via ELISA assay.
Changes in plasma Transforming Growth Factor (TGF)-β level | Baseline, 12 weeks
  TGF-β level will be assessed in plasma samples via ELISA assay.
Changes in ROS production capacity | Baseline, 12 weeks
  ROS production will be evaluated by the superoxide dismutase-sensitive cytochrome C reduction assay and results of these assays will be expressed as nmol of reduced cytochrome C / 10^6 cells / 30 min.

SECONDARY OUTCOMES:
Changes in Naive-Memory lymphocytes subpopulations | Baseline, 12 weeks
  Lymphocytes subpopulations will be assessed through flow cytometry with panel Naive-Mem + CD45V500 (CD45/CD3/CD4/CD8/CD45RA/CCR7).
  The following subpopulations will be assessed as percentage of parent population: CD3+ lymphocytes (% of ly CD45+), CD4+ T lymphocytes (% of CD3+) CD4+ T Naive (% of CD4+), CD4+ T Central Memory (CM) (% of CD4+), CD4+ T Effector Memory (EM), (% of CD4+), CD4+ T Effector Memory cells Re-expressing CD45RA (EMRA) (% of CD4+).
Changes in T helper (Th) lymphocytes subpopulations | Baseline, 12 weeks
  Lymphocytes subpopulations will be assessed through flow cytometry with panel Th+CD3+CD45V500 (CD45/CD3/CD4/CXCR3/CCR4/CCR6).
  The following subpopulations will be assessed as percentage of parent population: CD3+ lymphocytes (% of lyCD45+), CD4+ T lymphocytes (% of CD3+), Th1 (% of CD4+), Th1-Th17 (% of CD4+), Th2 (% of CD4+), Th17 (% of CD4+).
Changes in Regulatory T cells (Treg) lymphocytes subpopulations | Baseline, 12 weeks
  Lymphocytes subpopulations will be assessed through flow cytometry with panel TREG+CD3+CD45V500 (CD45/CD3/CD4/CD25/CD127/CD45RA).
  The following subpopulations will be assessed as percentage of parent population: CD3+ lymphocytes (% Ly CD45+), CD4+ T lymphocytes (% of CD3+), CD4+ Treg (% of CD4+), Naïve Treg (% of Treg), Active Treg (% of Treg).
Changes in Monocyte subpopulations | Baseline, 12 weeks
  Monocytes subpopulations will be assessed through flow cytometry with Monocyte Panel (CD45/HLA-DR/CD14/CD16).
  The following subpopulations will be assessed as percentage of parent population: Classical Monocytes (% of all HLA-DR+ Monocytes), Intermediate Monocytes (% of all HLA-DR+ Monocytes), Non-Classical Monocytes (% of all HLA-DR+ Monocytes).
  The three assessed subsets will also be characterised by their Median Fluorescence Intensity (MFI).
Changes in NK subpopulations | Baseline, 12 weeks
  NK cells subpopulations will be assessed through flow cytometry with NK-NKT Cell Panel (CD45/CD3/CD56/CD16/CD57/CD14/CD19).
  The following subpopulations will be assessed as percentage of parent population: NK cells (% of Ly CD45+), CD56dim/CD16bright (% of NK), CD56bright/CD16dim (% of NK), CD57- (% of CD56dim/CD16bright), CD57+ (% of CD56dim/CD16bright), CD57- (% of CD56bright/CD16dim), CD57+ (% of CD56bright/CD16dim).
Changes in CD4+ T cells TBX21 mRNA levels | Baseline, 12 weeks
  mRNA levels of the transcription factor gene TBX21 will be assessed through RT-PCR
Changes in CD4+ T cells STAT1 mRNA levels | Baseline, 12 weeks
  mRNA levels of the transcription factor gene STAT1 will be assessed through RT-PCR
Changes in CD4+ T cells STAT3 mRNA levels | Baseline, 12 weeks
  mRNA levels of the transcription factor gene STAT3 will be assessed through RT-PCR
Changes in CD4+ T cells STAT4 mRNA levels | Baseline, 12 weeks
  mRNA levels of the transcription factor gene STAT4 will be assessed through RT-PCR
Changes in CD4+ T cells STAT6 mRNA levels | Baseline, 12 weeks
  mRNA levels of the transcription factor gene STAT6 will be assessed through RT-PCR
Changes in CD4+ T cells RORC mRNA levels | Baseline, 12 weeks
  mRNA levels of the transcription factor gene RORC will be assessed through RT-PCR
Changes in CD4+ T cells GATA3 mRNA levels | Baseline, 12 weeks
  mRNA levels of the transcription factor gene GATA3 will be assessed through RT-PCR
Changes in CD4+ T cells FOXP3 mRNA levels | Baseline, 12 weeks
  mRNA levels of the transcription factor gene FOXP3 will be assessed through RT-PCR
Changes in CD4+ T cells NR4A2 mRNA levels | Baseline, 12 weeks
  mRNA levels of the transcription factor gene NR4A2 will be assessed through RT-PCR

OTHER OUTCOMES:
Changes in Unified Parkinson's Disease Rating Scale (UPDRS) scores | Baseline, 6 weeks, 12 weeks
  Scores for the UPDRS will be collected for all participants during scheduled visits.
  Minimum score is 0 and maximum score is 199, with higher scores representing worse outcomes.
Changes in Hoehn and Yahr's (H&Y) assessment scale | Baseline, 6 weeks, 12 weeks
  Scores for the H&Y assessment will be collected for all participants during scheduled visits.
  H&Y scale includes stages from 0 to 5. Intermediate stages 1.5 and 2.5 are widely used. A higher stage represents worse clinical conditions.
Changes in Non-Motor Symptoms Scale in Parkinson's disease (NMSS) scores | Baseline, 6 weeks, 12 weeks
  Scores for the NMSS will be collected for all participants during scheduled visits.
  The NMSS is divided into 9 different domains and 30 single questions on non-motor symptoms severity and frequency. Severity is reported from 0 (None) to 3 (Severe), frequency is can range from 1 (Rarely) to 4 (Very Frequent). Each question yields a Frequency x Severity value and total minimum score is 0, while maximum is 360. Higher scores represent more frequent and more severe non-motor symptoms.
Changes in Beck's Depression Inventory Scale (BDI-II) scores | Baseline, 6 weeks, 12 weeks
  Scores for BDI-II will be collected for all participants during scheduled visits.
  BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
  Minimum score is 0 and maximum score is 63.
Changes in Zung's Self Rating Anxiety Scale (SAS) scores | Baseline, 6 weeks, 12 weeks
  Scores for SAS will be collected for all participants during scheduled visits. This scale consists of 20 statements for which a frequency self-assessment is requested.
  Minimum score is 20, maximum score is 80, with higher scores representing worse anxiety symptoms.
Changes in Composite Autonomic Symptoms Scale 31 (COMPASS-31) scores | Baseline, 6 weeks, 12 weeks
  Scores for COMPASS-31 will be collected for all participants during scheduled visits.
  COMPASS-31 total scores can range between 0 to 100, with higher values representing more severe symptoms.
Changes in Montreal Cognitive Assessment (MOCA) scores | Baseline, 6 weeks, 12 weeks
  Scores for MOCA will be collected for all participants during scheduled visits. Total scores for MOCA range between 0 and 30, with lower scores representing worse cognitive performance.
Changes in the Patient Assessment of Constipation - Quality Of Life (PAC-QOL) questionnaire | Baseline, 6 weeks, 12 weeks
  Scores for PAC-QOL will be collected for all participants during scheduled visits.
  The range of possible scores on this questionnaire is 0 to 112, with higher scores indicative of a greater burden of constipation on quality of life.
Changes in reported Bristol Stool Form Chart assessment | Baseline, 6 weeks, 12 weeks
  Bristol Stool Form Chart will be used upon scheduled visits to evaluate stool form changes.
  This data is qualitative and values are not representative per se of better or worse outcomes or symptoms.
Changes in Constipation Assessment Scale (CAS) scores | Baseline, 6 weeks, 12 weeks
  Scores for CAS will be collected for all participants during scheduled visits. CAS scores range from 0 to 16 and are calculated on 8 items rated from 0 (no problem) to 2 (severe problem). Higher scores represent worse constipation symptoms.
Changes in Wexner Constipation Scoring System (WCSS) scores | Baseline, 6 weeks, 12 weeks
  Scores for WCSS will be collected for all participants during scheduled visits. Possible values for the WCSS range from 0 to 30, with higher scores representing worse constipation symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Franca Marino, Prof., Principal Investigator — Centre for Research in Medical Pharmacology
Locations (1):
- Azienda Ospedaliero-Universitaria "Maggiore della Carità", Novara, Italy

IPD SHARING:
Plan to Share IPD: Yes
All data collected during the trial, in anonymised form, will be made available to other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication of the final results.
Access Criteria: Requests to access collected data will be reviewed by academic staff at the Centre for Research in Medical Pharmacology, where all data will be stored. Access will be granted to researchers and clinical staff sharing a documented outline of their intended project.

REFERENCES:
- [Background] Tysnes OB, Storstein A. Epidemiology of Parkinson's disease. J Neural Transm (Vienna). 2017 Aug;124(8):901-905. doi: 10.1007/s00702-017-1686-y. Epub 2017 Feb 1. PMID 28150045
- [Background] Armstrong MJ, Okun MS. Diagnosis and Treatment of Parkinson Disease: A Review. JAMA. 2020 Feb 11;323(6):548-560. doi: 10.1001/jama.2019.22360. PMID 32044947
- [Background] Stefanis L. alpha-Synuclein in Parkinson's disease. Cold Spring Harb Perspect Med. 2012 Feb;2(2):a009399. doi: 10.1101/cshperspect.a009399. PMID 22355802
- [Background] Comi C, Tondo G. Insights into the protective role of immunity in neurodegenerative disease. Neural Regen Res. 2017 Jan;12(1):64-65. doi: 10.4103/1673-5374.198980. No abstract available. PMID 28250745
- [Background] Cappellano G, Carecchio M, Fleetwood T, Magistrelli L, Cantello R, Dianzani U, Comi C. Immunity and inflammation in neurodegenerative diseases. Am J Neurodegener Dis. 2013 Jun 21;2(2):89-107. Print 2013. PMID 23844334
- [Background] Liu X, Yamada N, Maruyama W, Osawa T. Formation of dopamine adducts derived from brain polyunsaturated fatty acids: mechanism for Parkinson disease. J Biol Chem. 2008 Dec 12;283(50):34887-95. doi: 10.1074/jbc.M805682200. Epub 2008 Oct 15. PMID 18922792
- [Background] Kustrimovic N, Rasini E, Legnaro M, Bombelli R, Aleksic I, Blandini F, Comi C, Mauri M, Minafra B, Riboldazzi G, Sanchez-Guajardo V, Marino F, Cosentino M. Dopaminergic Receptors on CD4+ T Naive and Memory Lymphocytes Correlate with Motor Impairment in Patients with Parkinson's Disease. Sci Rep. 2016 Sep 22;6:33738. doi: 10.1038/srep33738. PMID 27652978
- [Background] Kustrimovic N, Comi C, Magistrelli L, Rasini E, Legnaro M, Bombelli R, Aleksic I, Blandini F, Minafra B, Riboldazzi G, Sturchio A, Mauri M, Bono G, Marino F, Cosentino M. Parkinson's disease patients have a complex phenotypic and functional Th1 bias: cross-sectional studies of CD4+ Th1/Th2/T17 and Treg in drug-naive and drug-treated patients. J Neuroinflammation. 2018 Jul 12;15(1):205. doi: 10.1186/s12974-018-1248-8. PMID 30001736
- [Background] De Francesco E, Terzaghi M, Storelli E, Magistrelli L, Comi C, Legnaro M, Mauri M, Marino F, Versino M, Cosentino M. CD4+ T-cell Transcription Factors in Idiopathic REM Sleep Behavior Disorder and Parkinson's Disease. Mov Disord. 2021 Jan;36(1):225-229. doi: 10.1002/mds.28137. Epub 2020 Jul 10. PMID 32649001
- [Background] Tekriwal A, Kern DS, Tsai J, Ince NF, Wu J, Thompson JA, Abosch A. REM sleep behaviour disorder: prodromal and mechanistic insights for Parkinson's disease. J Neurol Neurosurg Psychiatry. 2017 May;88(5):445-451. doi: 10.1136/jnnp-2016-314471. Epub 2016 Dec 13. PMID 27965397
- [Background] Cersosimo MG, Raina GB, Pecci C, Pellene A, Calandra CR, Gutierrez C, Micheli FE, Benarroch EE. Gastrointestinal manifestations in Parkinson's disease: prevalence and occurrence before motor symptoms. J Neurol. 2013 May;260(5):1332-8. doi: 10.1007/s00415-012-6801-2. Epub 2012 Dec 21. PMID 23263478
- [Background] Comi C, Magistrelli L, Oggioni GD, Carecchio M, Fleetwood T, Cantello R, Mancini F, Antonini A. Peripheral nervous system involvement in Parkinson's disease: evidence and controversies. Parkinsonism Relat Disord. 2014 Dec;20(12):1329-34. doi: 10.1016/j.parkreldis.2014.10.010. Epub 2014 Oct 18. PMID 25457816
- [Background] McCann H, Cartwright H, Halliday GM. Neuropathology of alpha-synuclein propagation and braak hypothesis. Mov Disord. 2016 Feb;31(2):152-60. doi: 10.1002/mds.26421. Epub 2015 Sep 4. PMID 26340605
- [Background] Sampson TR, Debelius JW, Thron T, Janssen S, Shastri GG, Ilhan ZE, Challis C, Schretter CE, Rocha S, Gradinaru V, Chesselet MF, Keshavarzian A, Shannon KM, Krajmalnik-Brown R, Wittung-Stafshede P, Knight R, Mazmanian SK. Gut Microbiota Regulate Motor Deficits and Neuroinflammation in a Model of Parkinson's Disease. Cell. 2016 Dec 1;167(6):1469-1480.e12. doi: 10.1016/j.cell.2016.11.018. PMID 27912057
- [Background] Magistrelli L, Amoruso A, Mogna L, Graziano T, Cantello R, Pane M, Comi C. Probiotics May Have Beneficial Effects in Parkinson's Disease: In vitro Evidence. Front Immunol. 2019 May 7;10:969. doi: 10.3389/fimmu.2019.00969. eCollection 2019. PMID 31134068
- [Background] Tankou SK, Regev K, Healy BC, Cox LM, Tjon E, Kivisakk P, Vanande IP, Cook S, Gandhi R, Glanz B, Stankiewicz J, Weiner HL. Investigation of probiotics in multiple sclerosis. Mult Scler. 2018 Jan;24(1):58-63. doi: 10.1177/1352458517737390. PMID 29307299
- [Background] Tankou SK, Regev K, Healy BC, Tjon E, Laghi L, Cox LM, Kivisakk P, Pierre IV, Hrishikesh L, Gandhi R, Cook S, Glanz B, Stankiewicz J, Weiner HL. A probiotic modulates the microbiome and immunity in multiple sclerosis. Ann Neurol. 2018 Jun;83(6):1147-1161. doi: 10.1002/ana.25244. Epub 2018 Jun 8. PMID 29679417
- [Background] Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. The Unified Parkinson's Disease Rating Scale (UPDRS): status and recommendations. Mov Disord. 2003 Jul;18(7):738-50. doi: 10.1002/mds.10473. PMID 12815652
- [Background] Goetz CG, Poewe W, Rascol O, Sampaio C, Stebbins GT, Counsell C, Giladi N, Holloway RG, Moore CG, Wenning GK, Yahr MD, Seidl L; Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. Movement Disorder Society Task Force report on the Hoehn and Yahr staging scale: status and recommendations. Mov Disord. 2004 Sep;19(9):1020-8. doi: 10.1002/mds.20213. PMID 15372591
- [Background] van Wamelen DJ, Martinez-Martin P, Weintraub D, Schrag A, Antonini A, Falup-Pecurariu C, Odin P, Ray Chaudhuri K; International Parkinson and Movement Disorder Society Parkinson's Disease Non-Motor Study Group. The Non-Motor Symptoms Scale in Parkinson's disease: Validation and use. Acta Neurol Scand. 2021 Jan;143(1):3-12. doi: 10.1111/ane.13336. Epub 2020 Sep 29. PMID 32813911
- [Background] Visser M, Leentjens AF, Marinus J, Stiggelbout AM, van Hilten JJ. Reliability and validity of the Beck depression inventory in patients with Parkinson's disease. Mov Disord. 2006 May;21(5):668-72. doi: 10.1002/mds.20792. PMID 16450355
- [Background] Dunstan DA, Scott N. Norms for Zung's Self-rating Anxiety Scale. BMC Psychiatry. 2020 Feb 28;20(1):90. doi: 10.1186/s12888-019-2427-6. PMID 32111187
- [Background] Zung WW. A rating instrument for anxiety disorders. Psychosomatics. 1971 Nov-Dec;12(6):371-9. doi: 10.1016/S0033-3182(71)71479-0. No abstract available. PMID 5172928
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] Kim Y, Seok JM, Park J, Kim KH, Min JH, Cho JW, Park S, Kim HJ, Kim BJ, Youn J. The composite autonomic symptom scale 31 is a useful screening tool for patients with Parkinsonism. PLoS One. 2017 Jul 6;12(7):e0180744. doi: 10.1371/journal.pone.0180744. eCollection 2017. PMID 28683089
- [Background] Vasquez KA, Valverde EM, Aguilar DV, Gabarain HH. Montreal Cognitive Assessment scale in patients with Parkinson Disease with normal scores in the Mini-Mental State Examination. Dement Neuropsychol. 2019 Jan-Mar;13(1):78-81. doi: 10.1590/1980-57642018dn13-010008. PMID 31073382
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Background] Dal Molin A, McMillan SC, Zenerino F, Rattone V, Grubich S, Guazzini A, Rasero L. Validity and reliability of the Italian Constipation Assessment Scale. Int J Palliat Nurs. 2012 Jul;18(7):321-5. doi: 10.12968/ijpn.2012.18.7.321. PMID 22885963
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] Del Piano M, Carmagnola S, Anderloni A, Andorno S, Ballare M, Balzarini M, Montino F, Orsello M, Pagliarulo M, Sartori M, Tari R, Sforza F, Capurso L. The use of probiotics in healthy volunteers with evacuation disorders and hard stools: a double-blind, randomized, placebo-controlled study. J Clin Gastroenterol. 2010 Sep;44 Suppl 1:S30-4. doi: 10.1097/MCG.0b013e3181ee31c3. PMID 20697291
- [Background] Chng KR, Ghosh TS, Tan YH, Nandi T, Lee IR, Ng AHQ, Li C, Ravikrishnan A, Lim KM, Lye D, Barkham T, Raman K, Chen SL, Chai L, Young B, Gan YH, Nagarajan N. Metagenome-wide association analysis identifies microbial determinants of post-antibiotic ecological recovery in the gut. Nat Ecol Evol. 2020 Sep;4(9):1256-1267. doi: 10.1038/s41559-020-1236-0. Epub 2020 Jul 6. PMID 32632261
- [Background] Duranti S, Ruiz L, Lugli GA, Tames H, Milani C, Mancabelli L, Mancino W, Longhi G, Carnevali L, Sgoifo A, Margolles A, Ventura M, Ruas-Madiedo P, Turroni F. Bifidobacterium adolescentis as a key member of the human gut microbiota in the production of GABA. Sci Rep. 2020 Aug 24;10(1):14112. doi: 10.1038/s41598-020-70986-z. PMID 32839473
- [Background] Kimmelman J, Mogil JS, Dirnagl U. Distinguishing between exploratory and confirmatory preclinical research will improve translation. PLoS Biol. 2014 May 20;12(5):e1001863. doi: 10.1371/journal.pbio.1001863. eCollection 2014 May. PMID 24844265
- [Derived] Martini S, Marino F, Magistrelli L, Contaldi E, Cosentino M, Comi C. The PROB-PD trial: a pilot, randomised, placebo-controlled study protocol to evaluate the feasibility and potential efficacy of probiotics in modulating peripheral immunity in subjects with Parkinson's disease. Pilot Feasibility Stud. 2023 May 8;9(1):77. doi: 10.1186/s40814-023-01306-1. PMID 37158925